CLINICAL TRIAL: NCT01033344
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate Two Treatment Regimens of Cat-PAD in Cat Allergic Subjects Following Challenge to Cat Allergen in an Environmental Exposure Chamber
Brief Title: Cat-PAD Exposure Chamber Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry); Cetero Research, San Antonio (Network)
Responsible Party: Dr Rod Hafner, Circassia Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP005
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Cat Allergy
Keywords: Cat allergy; Rhinoconjunctivitis; Exposure chamber; Immunotherapy; Cat-PAD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Solution resembling active solution but without peptides
  Interventions: Biological: Placebo
- Group 1 (Experimental): Cat-PAD dose group 1
  Interventions: Biological: Cat-PAD
- Group 2 (Experimental): Cat-PAD Dose group 2
  Interventions: Biological: Cat-PAD

INTERVENTIONS:
Biological: Placebo — Intradermal injection 1x8 administrations 2 weeks apart
  Arms: Placebo
Biological: Cat-PAD — Intradermal injection 1x8 administrations 2 weeks apart
  Arms: Group 1
Biological: Cat-PAD — Intradermal injection, 1x8 administrations 2 weeks apart, alternating active and placebo
  Arms: Group 2

SUMMARY:
Cat allergy is an increasingly prevalent condition, affecting 10-15% of patients with allergic rhinoconjunctivitis and/or asthma. Cat-PAD is a novel, synthetic, allergen-derived peptide desensitising vaccine, currently being developed for the treatment of cat allergy.

This study will look at the efficacy, safety and tolerability of two doses of Cat-PAD in cat allergic subjects following challenge to cat allergen in an EEC.

DETAILED DESCRIPTION:
This study is designed as a randomised, double-blind, placebo-controlled, parallel group study to evaluate the safety and tolerability of Cat-PAD in cat allergic subjects with allergic rhinoconjunctivitis,subjects may also have controlled asthma. The efficacy of Cat-PAD will be explored in subjects using an(Environmental Exposure Chamber)EEC.

The study will consist of 3 study periods. In Period 1, Screening will be performed up to a maximum of 12 weeks before randomisation and may consist of one or two visits to the clinic, at the Investigator's discretion. Baseline Challenge will consist of 4 visits to the EEC at least 3 days before randomisation.

In Period 2, subjects in each cohort complying with the inclusion/exclusion criteria will be randomised to one of three groups and will receive treatment every 2 weeks (±2 days) for 14 weeks.

In Period 3, Post Treatment Challenge will consist of 4 visits to the EEC 18-22 weeks after the first administration in the treatment period and assessments will be performed identical to those at the baseline challenge. Follow-up will be conducted 3-10 days after PTC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years
* Minimum 1-year history of rhinoconjunctivitis on exposure to cats. (Subjects may also have controlled asthma)
* Positive skin prick test to cat allergen with a wheal diameter at least 3mm larger than that produced by the negative control
* Minimum qualifying rhinoconjunctivitis symptom scores

Exclusion Criteria:

* "Partly controlled" and "uncontrolled" asthma
* History of anaphylaxis to cat allergen
* FEV1 of less than 70% of predicted
* Subjects who cannot tolerate baseline challenge in the EEC
* Treatment with beta-blockers,Alpha-adrenoceptor blockers, Tranquillizers or psychoactive drugs
* A history of any significant disease or disorder (e.g. cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, neoplastic/malignant, psychiatric, major physical impairment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Total Rhinoconjunctivitis Symptom Score | 0 and 18-22 weeks after start of treatment

SECONDARY OUTCOMES:
Symptom scores for ocular and nasal symptoms | 0 and 18-22 weeks after start of treatment
Acoustic Rhinometry | 0 and 18-22 weeks after start of treatment
Cat Specific IgE | At 0 weeks and at follow up
Adverse Events | During study

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, CCF, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Mississauga, Ontario, Canada